CLINICAL TRIAL: NCT06664359
Title: Avoid Pneumothorax: Identification of the Interscapular Area Trigger Point Injection Safe Zone in Different Positions (Sitting/Prone)
Brief Title: Safe Zone in Trigger Point Injection
Status: Recruiting | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Süheyla Karadağ Erkoç, Medical Doctor, Ankara University
Other Study IDs: 2024/376
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Trigger Point Pain, Myofascial
Keywords: Trigger Point Pain; Myofascial pain; ultrasound; pneumothorax
MeSH Terms: conditions — Myofascial Pain Syndromes; Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- myofascial pain: myofascial pain syndrome
  Interventions: Other: Ultrasound guided injection with local anaestethic

INTERVENTIONS:
Other: Ultrasound guided injection with local anaestethic — Volunteers will first be asked to sit on a chair with their back facing the examiner, placing their arms in a relaxed position with their head supported on a surface in front of them. The ultrasound operator will be positioned behind the volunteer. Initially, in the sitting position, volunteers will be asked to maintain normal breathing. Once an optimal ultrasound image is obtained, the image will be frozen, and measurements will be taken from the same image in sequence. The measurements to be performed are as follows: skin-fat tissue distance, skin-trapezius muscle distance, skin-rhomboid muscle distance, skin-rib distance, skin-pleura distance, and rhomboid muscle-pleura distance. These measurements, in millimeters, will be recorded in the data collection form. The same measurements will also be taken during deep inhalation and deep exhalation in the sitting position."
Other: Ultrasound guided injection with local anaestethic — Volunteers will first be asked to lay prone position.The ultrasound operator will be positioned behind the volunteer. Initially, in the sitting position, volunteers will be asked to maintain normal breathing. Once an optimal ultrasound image is obtained, the image will be frozen, and measurements will be taken from the same image in sequence. The measurements to be performed are as follows: skin-fat tissue distance, skin-trapezius muscle distance, skin-rhomboid muscle distance, skin-rib distance, skin-pleura distance, and rhomboid muscle-pleura distance. These measurements, in millimeters, will be recorded in the data collection form. The same measurements will also be taken during deep inhalation and deep exhalation in the sitting position."

SUMMARY:
The goal of this observational study is to define the safe distance that will reduce the risk of pneumothorax through ultrasonographic imaging measurements in both sitting and prone positions to ensure patient safety during these procedures. The main question[s] it aims to answer [is/are]:

The mean distance between the skin and pleura in sitting position during the inhalation and exhalation The mean distance between the skin and pleura in prone position during the inhalation and exhalation

DETAILED DESCRIPTION:
Myofascial pain syndrome is characterized by pain and tenderness at specific points known as trigger points. Tension and spasm occur in the muscles, making it one of the most common causes of musculoskeletal pain. Various treatment options, such as TENS, dry needling, and trigger point injections, are available for the management of myofascial pain syndrome. Trigger point injection is one of the evidence based treatment methods that can provide both temporary and long-term relief.

Trigger point injections can be performed under ultrasound guidance or by blind technique. Although trigger point injection is generally be considered a safe procedure when performed by a skilled practitioner, complications may occur. These complications include pain during and after the procedure, nerve injury, bleeding, infection, and serious complications such as pneumothorax. Pneumothorax may occur when trigger point injections are administered into the chest wall muscles, particularly the trapezius, rhomboid major, or rhomboid minor muscles. Among these muscles, the rhomboid major is very thin, and the thickness of the skin, subcutaneous fat layer, and other soft tissues surrounding it varies between individuals. Since nerves, vascular structures, and the pleura are present in the deeper parts of these muscles, determining the appropriate injection depth is crucial.

In clinical practice, trigger point injections are administered by clinicians in both prone and sitting positions. To the best of our knowledge there is no studies thatinvestigates the determination of a safe distance through measurements in both the sitting and prone positions. In this study we aim to calculate the safe distance using ultrasound that will reduce the risk of pneumothorax through ultrasonographic imaging measurements in both sitting and prone positions during inhalation and exhalation to ensure patient safety during these procedures.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with Myofascial Pain Syndrome
* patients scheduled for trigger point injections due to Myofascial Pain Syndrome.

Exclusion Criteria:

* under 18 years of age,
* additional diseases other than Myofascial Pain Syndrome,
* the presence of active infection in the interscapular area where ultrasound imaging and measurements will be performed,
* lesions that disrupt skin integrity or affect subcutaneous and muscle structures such as anomalies or masses that could impair imaging quality
* individuals with known lung diseases
* not consent to participate in the study."

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo trigger point injections due to myofascial pain
Sampling Method: Non-Probability Sample
Enrollment: 211 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
skin-pleura distance in sitting position | 1 day
  Evaluate the skin-pleura distance in sitting position during inhalation and exhalation
skin-pleura distance in prone position | 1 day
  skin-pleura distance in prone position during inhalation and exhalation

SECONDARY OUTCOMES:
the correlation of skin-pleura distance and body mass index | 1 day
  the correlation of skin-pleura distance in sitting and prone position and body mass index
the correlation of skin-pleura distance and dominant hand | 1 day
  the correlation of skin-pleura distance in sitting and prone position and dominant hand
the correlation of skin-pleura distance and the chest wall diameter | 1 day
  the correlation of skin-pleura distance in sitting and prone position and the chest wall diameter

CONTACTS AND LOCATIONS:
Overall Officials: Suheyla Karadağ-Erkoç, MD, Study Director — Department of Anesthesiology and Reanimation, Ankara University, Ankara, Turkey
Locations (1):
- Ankara University Department of Anesthesiology and Reanimation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mitchell UH, Johnson AW, Larson RE, Seamons CT. Positional changes in distance to the pleura and in muscle thickness for dry needling. Physiotherapy. 2019 Sep;105(3):362-369. doi: 10.1016/j.physio.2018.08.002. Epub 2018 Aug 18. PMID 30343872